CLINICAL TRIAL: NCT00018226
Title: Enhanced Outreach Counseling Following Methadone Treatment Discharge
Brief Title: Effect Of Case Management Following Discharge From Methadone Treatment
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: US Department of Veterans Affairs (U.S. Federal Agency)
Organization: VA Office of Research and Development (U.S. Federal Agency)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ADRD-022-97S
Record Dates: First submitted 2001-07-03; First posted 2001-07-05 (Estimated); Last update posted 2009-01-21 (Estimated); Status verified 2004-12

CONDITIONS: Opioid-Related Disorders
MeSH Terms: conditions — Opioid-Related Disorders | interventions — Case Management

INTERVENTIONS:
Behavioral: Case Management

SUMMARY:
The purpose of this project is to assess whether enhanced outreach counseling (EOC) is an effective outreach strategy for discharged methadone maintenance patients compared to a standard referral procedure. EOC is a brief (30 minute) face-to-face intervention, followed by six weeks of ongoing telephone counseling/case management designed to help eligible out-of-treatment methadone patients re-enter treatment. Several studies have shown those patients who voluntarily re-enter treatment improve significantly following re-enrollment.

ELIGIBILITY:
Patients who have been discharged from methadone maintenance treatment at the PVAMC who consented (as active patients) to be contacted for follow-up upon discharge.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 1998-04; Study Completion 2001-03

CONTACTS AND LOCATIONS:
Locations (1):
- Drug Dependent Treatment Unit, Philadelphia, Pennsylvania, United States